CLINICAL TRIAL: NCT04953039
Title: Use of Saliva for Diagnosis of SARS-CoV2 Infection
Brief Title: Use of Saliva for COVID-19 Diagnosis
Acronym: SALIVA-01
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Giorgio Novelli, Principal Investigator, University of Milano Bicocca
Other Study IDs: SALIVA-01
Record Dates: First submitted 2021-06-08; First posted 2021-07-07 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV2 Infection
Keywords: Salivary test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to evaluate the presence of SARS-CoV2 RNA in the saliva of patients with suspected or confirmed COVID-19 in order to validate the analysis of this type of sample for the diagnosis of SARS-CoV2 infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age hospitalized in the COVID-19 wards of ASST Monza - San Gerardo Hospital with positive, weakly positive or negative nasopharyngeal swabs; initially assessed at the E.R.; symptomatic or asymptomatic with indication to hospitalization.
* Informed consent freely granted and acquired before the start of the study.

Exclusion Criteria:

* Patients with significant clinical conditions which could interfere with the study in the opinion of the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed SARS-CoV2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Presence of SARS-CoV2 RNA in the saliva of patient with suspected or confirmed COVID-19. | Up to 52 weeks
  Positive - Negative

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Novelli, MD, Principal Investigator — ASST Monza - Ospedale San Gerardo
Locations (1):
- ASST MONZA - Ospedale San Gerardo, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided